CLINICAL TRIAL: NCT03679104
Title: Endoscopic Clips Versus Overstich Suturing System Device for Closure of Mucosotomy After Per-oral Endoscopic Pyloromyotomy (G-POEM)
Brief Title: Endoscopic Clips Versus Overstich Suturing System Device for Closure of Mucosotomy After G-POEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Doc. (Ass. prof.) Jan Martinek, MD, PhD, AGAF, Ass. prof., Institute for Clinical and Experimental Medicine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IClinicalEM3
Record Dates: First submitted 2018-08-12; First posted 2018-09-20 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Gastroparesis
Keywords: Gastric Per-oral Endoscopic Pyloromyotomy
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Intervention Model Description: Patients will be allocated to the corresponding group according to a peri-procedural finding, availability of a respective closure method and endoscopist´s decision.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic clips (Active Comparator): Closure of mucosotomy using endoscopic clips
  Interventions: Procedure: Closure of mucosotomy using endoscopic clips
- OverStitch™ suturing device (Active Comparator): Closure of mucosotomy using OverStitch™ suturing device
  Interventions: Procedure: Closure of mucosotomy using OverStitch™ suturing device

INTERVENTIONS:
Procedure: Closure of mucosotomy using endoscopic clips — Gastric per-oral endoscopic pyloromyotomy procedure requires the incision in the mucosa and submucosa. The closure of this incision at the end of the procedure will be done using endoscopic clips. These are used in endoscopy to mechanically close two mucosal surfaces without the need for surgery and suturing. In this study, the following endoclips may be used: Resolution 360™ Clip (Boston Scientific), QuickClip Pro™(Olympus) or Instinct™ Endoscopic Hemoclip (Cook Medical).
  Arms: Endoscopic clips
Procedure: Closure of mucosotomy using OverStitch™ suturing device — Gastric per-oral endoscopic pyloromyotomy procedure requires the incision in the mucosa and submucosa. The closure of this incision at the end of the procedure will be done by OverStitch™ (Apollo Endosurgery Inc., Austin, Texas, USA), which is a suturing device that enables advanced endoscopic surgery by allowing physicians to place full-thickness sutures through a flexible endoscope.
  Arms: OverStitch™ suturing device

SUMMARY:
Gastric per-oral endoscopic pyloromyotomy (G-POEM) has been assessed as new modality for treatment of refractory gastroparesis. G-POEM is promising method, which is still under investigation as its safety and efficacy has not been established yet. The ideal closure technique in patients undergoing G-POEM needs to be established. Several techniques may be used for endoscopic mucosal closure: endoscopic clips, OTSC (over the scope clips), endo-loop based methods (KING closure) or endoscopic suture.

The aim of this prospective, open-label study is to compare efficacy and safety of two methods for incision closure in patients who undergo G-POEM: endoscopic clips vs. endoscopic suturing system (OverStitch).

DETAILED DESCRIPTION:
Based on principles of NOTES (natural orifice transluminal endoscopic surgery), a mini-invasive therapeutic procedure such as per-oral endoscopic myotomy (POEM) or gastric per-oral endoscopic pyloromyotomy (G-POEM) have been assessed as new modalities for treatment of oesophageal achalasia or refractory gastroparesis. G-POEM is a new and promising method, which is still under investigation as its safety and efficacy has not been established yet. There are several questions, which need to be answered before G-POEM is considered as a standard clinical procedure. These questions concern, among others, efficacy, safety, technical performance etc. Mucosal incision should be endoscopically closed to prevent leakage into the abdominal cavity. Obtaining adequate mucosal closure is one of the most important steps of the procedure and is essential in avoiding major morbidity. The ideal closure technique in patients undergoing G-POEM needs to be established. Several techniques may be used for endoscopic mucosal closure: endoscopic clips, OTSC clips, endo-loop based methods (KING closure) or endoscopic suture. At present, simple closure with endoscopic clips has been the most frequently described method for mucosal closure in patients undergoing G-POEM. However, as gastric mucosa is thicker compared to the esophagus, where clips are used for POEM without any major problems, several authors have described problems during gastric incision closure - it takes a rather longer time, some clips cannot be placed and in some patients, other closure method had to be used. Thus, endoscopic clips may not be an ideal closure method in the stomach. A platform that replicates a principle of surgical suturing is endoscopic suturing system.

The aim of this prospective, open-label study is to compare efficacy and safety of two methods for incision closure in patients who undergo G-POEM: endoscopic clips vs. endoscopic suturing system (OverStitch).

Investigators plan to randomize 30-40 patients (15-20 in both arms, ratio 1:1).

The assigned closure method will be decided by an endoscopist prior to starting closure.

ELIGIBILITY:
Inclusion Criteria:

1. Refractory (> 6 months) and severe (based on a validated total Gastroparesis Cardinal Symptom Index) gastroparesis, with confirmed gastric emptying based on a gastric emptying study: standardized protocol of scintigraphy in all patients (performed less than 6 months prior to enrolment). The total GSCI (Gastroparesis Cardinal Symptom Index) score must be >2.0

   * Abnormal gastric emptying is defined as retention of Tc-99 m >60% at 2 h and/or ≥10% of residual activity at 4 h on a standardized sulphur colloid solid-phase gastric emptying study.
   * Abnormal gastric emptying breath test based on a solid normal range determination for the test used (e.g. T1/2 > 109 min)
2. Severe refractory disease is defined as GCSI >2.0 and failure or recurrence in patients who received available optimal pharmacological therapies.
3. Persons 18 years or older at the time of signing the informed consent
4. Signed informed consent

Exclusion Criteria:

1. No previous attempt with at least one prokinetic drug
2. No previous attempt to withdraw anticholinergic agents and glucagon like peptide -1 (GLP-1) and amylin analogues in patients treated with these substances
3. Active treatment with opioids or a history of treatment with opioids within 12 months before enrolment
4. Previous gastric surgery (Billroth I or Billroth II)
5. Known eosinophilic gastroenteritis
6. Organic pyloric (or intestinal) obstruction (fibrotic stricture, etc.)
7. Sever coagulopathy
8. Oesophageal or gastric varices and /or portal gastropathy
9. Advanced liver cirrhosis (Child B or Child C)
10. Active peptic ulcer disease
11. Pregnancy or puerperium
12. Malignant or pre-malignant gastric diseases (dysplasia, gastric cancer, GIST): patients with a history of such disease after its cure are eligible for enrolment
13. Any other condition, which in the opinion of the investigator would interfere with study requirements
14. Uncontrolled diabetes mellitus
15. Diagnosis of rumination syndrome or "eating" disorder (mental anorexia, bulimia nervosa)
16. Inability to obtain informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-01-26 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with successful and safe incision closure. | 3 months
  Definition of successful closure: endoscopically completely closed incision, no need to use another "rescue" closure method, no leak on post-operative day 1, no leak related complications, no readmission due to closure dehiscence, no need for surgery due to closure.

SECONDARY OUTCOMES:
Easiness of the closure | 3 months
  Handling with endoclips or OverStitch will be evaluated by means of a questionnaire where ease of use was scored on a VAS (visual analogue scale), 0 = impossible, 10 = very easy) by both, endoscopist as well as an endoscopy nurse assisting with the closure procedure.
Closure time of mucosotomy | 1 day
  The duration of endoscopic closure, reported by the endoscopist performing the procedure
Cost | 3 months
  To evaluate the economics and cost-effectiveness of treating gastroparesis
Healing quality | 3 months
  Assessing gastric scar after gastric per-oral pyloromyotomy: based on a visual examination, the healing process could include three stages, namely stage A (active stage): means no tissue reparation features, stage H (healing stage): early morphological reparation features, and stage S (scar stage): completed repair process, that could by described as S1 (red) or S2 (white). Width and length of scar will be measures as well.
Readmission within 30 days | 30 days
  A readmission for an endoscopic or surgery intervention to address a complication resulting from care during the initial admission.
Mortality at 3 months | 3 months
  Incidence of fatal complications related to procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jan Martinek, Study Chair — Department of Hepatogastroenterology, Institute for Clinical and Experimental Medicine, Prague, Czech Republic; Rastislav Hustak, Principal Investigator — Department of Hepatogastroenterology, Institute for Clinical and Experimental Medicine, Prague, Czech Republic; Zuzana Vackova, Principal Investigator — Department of Hepatogastroenterology, Institute for Clinical and Experimental Medicine, Prague, Czech Republic; Tomas Hucl, Principal Investigator — Department of Hepatogastroenterology, Institute for Clinical and Experimental Medicine, Prague, Czech Republic; Jan Usak, Principal Investigator — Universitary hospital Trnava, Slovak Republic; Julius Spicak, Prof, Principal Investigator — Department of Hepatogastroenterology, Institute for Clinical and Experimental Medicine, Prague, Czech Republic
Locations (1):
- Institute for Clinical and Experimental Medicine, Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Khashab MA, Ngamruengphong S, Carr-Locke D, Bapaye A, Benias PC, Serouya S, Dorwat S, Chaves DM, Artifon E, de Moura EG, Kumbhari V, Chavez YH, Bukhari M, Hajiyeva G, Ismail A, Chen YI, Chung H. Gastric per-oral endoscopic myotomy for refractory gastroparesis: results from the first multicenter study on endoscopic pyloromyotomy (with video). Gastrointest Endosc. 2017 Jan;85(1):123-128. doi: 10.1016/j.gie.2016.06.048. Epub 2016 Jun 25. PMID 27354102
- [Result] Dacha S, Mekaroonkamol P, Li L, Shahnavaz N, Sakaria S, Keilin S, Willingham F, Christie J, Cai Q. Outcomes and quality-of-life assessment after gastric per-oral endoscopic pyloromyotomy (with video). Gastrointest Endosc. 2017 Aug;86(2):282-289. doi: 10.1016/j.gie.2017.01.031. Epub 2017 Feb 1. PMID 28161449
- [Result] Paspatis GA, Dumonceau JM, Barthet M, Meisner S, Repici A, Saunders BP, Vezakis A, Gonzalez JM, Turino SY, Tsiamoulos ZP, Fockens P, Hassan C. Diagnosis and management of iatrogenic endoscopic perforations: European Society of Gastrointestinal Endoscopy (ESGE) Position Statement. Endoscopy. 2014 Aug;46(8):693-711. doi: 10.1055/s-0034-1377531. Epub 2014 Jul 21. PMID 25046348
- [Result] Kantsevoy SV, Bitner M, Mitrakov AA, Thuluvath PJ. Endoscopic suturing closure of large mucosal defects after endoscopic submucosal dissection is technically feasible, fast, and eliminates the need for hospitalization (with videos). Gastrointest Endosc. 2014 Mar;79(3):503-7. doi: 10.1016/j.gie.2013.10.051. Epub 2013 Dec 12. PMID 24332082
- [Result] Crichton NJ. Principles of statistical analysis in nursing and healthcare research. Nurse Res. 2001 Oct 1;9(1):4-16. doi: 10.7748/nr2001.10.9.1.4.c6171. PMID 26954377